CLINICAL TRIAL: NCT04985110
Title: Pemberian Antibiotik Profilaksis Pada Biopsi Prostat Transperineal di RSUPN Dr. Cipto Mangunkusumo: Uji Klinis Acak Terkontrol
Brief Title: Administration of Antibiotic Prophylaxis for Transperineal Prostate Biopsy in Cipto Mangunkusumo Hospital
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, dr. Agus Rizal Ardy Hariandy Hamid, Sp.U(K), Ph.D, Main Researcher, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 21-02-0154
Record Dates: First submitted 2021-07-26; First posted 2021-08-02 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-07

CONDITIONS: Prostate Cancer; Prostate Biopsy; Perioperative Complication; Bacteriuria; Urinary Tract Infections; Sepsis
Keywords: Antibiotic prophylaxis; Transperineal prostate biopsy; Randomized controlled trial
MeSH Terms: conditions — Prostatic Neoplasms; Bacteriuria; Urinary Tract Infections; Sepsis | interventions — Trimethoprim, Sulfamethoxazole Drug Combination

STUDY DESIGN:
Intervention Model Description: This randomized controlled trial aims to compare the rate of perioperative infection complications in transperineal prostate biopsy between the group that receives prophylactic antibiotic and the group that receives placebo.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The randomization process will be conducted before the study started. Computers will generate random numbers, which will put the participants into two groups. These numbers can only be accessed by the clinical research supporting unit team, while the investigators, surgeons, residents, nurses, and pharmacologists involved will be blinded to this information. To ensure patient blinding, the placebo will be manufactured as identical capsules.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cotrimoxazole (Experimental): The treatment group will receive Cotrimoxazole Forte 960 mg PO q.d. 4 hours before the biopsy procedure.
  Interventions: Drug: Cotrimoxazole
- Placebo (Placebo Comparator): The placebo group will receive placebo q.d. 4 hours before the biopsy procedure.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cotrimoxazole — The treatment group will receive Cotrimoxazole Forte 960 mg PO q.d. 4 hours before the biopsy procedure.
  Arms: Cotrimoxazole
Drug: Placebo — The placebo group will receive placebo q.d. 4 hours before the biopsy procedure.
  Arms: Placebo

SUMMARY:
This randomized controlled trial aims to compare the rate of perioperative infection complications in transperineal prostate biopsy between the group that receives prophylactic antibiotic and the group that receives placebo. The types of infection studied included bacteriuria, urinary tract infection (UTI), UTI with fever (febrile UTI), and sepsis. This study hypothesized that the administration of prophylactic antibiotics during transperineal prostate biopsy would result in lower rates of perioperative infection complications.

DETAILED DESCRIPTION:
Prostate cancer screenings will be conducted in all patients aged >45 years with lower urinary tract symptoms (LUTS) through PSA test and digital rectal examination (DRE). Those with PSA levels of 4.0 ng/mL or higher or other abnormal findings on DRE will be recommended to undergo transperineal prostate biopsy. In addition, participants will be offered to participate in this clinical trial, in which participants will be randomly assigned into two groups: one group will receive prophylactic antibiotic, while the other group will receive placebo.

The randomization process will be conducted before the biopsy procedure. Computers will generate random numbers, which will put the participants into two groups. These numbers can only be accessed by the research monitor (Clinical Research Supporting Unit of IMERI FMUI), while the investigators, surgeons, residents, and nurses involved will be blinded to this information. To ensure patient blinding, the placebo and cotrimoxazole forte 960 mg will be reformed as identical as possible in capsule preparation.

The primary outcomes of this clinical trial are the rate of perioperative infection complications, including bacteriuria, urinary tract infection (UTI), UTI with fever (febrile UTI), and sepsis, in 24 hours, 7 days, and 14 days postoperatively. The secondary outcomes of this clinical trial are the rate of readmission.

ELIGIBILITY:
Inclusion Criteria:

* Patient with lower urinary tract symptoms aged >45 years with either PSA levels of 4.0 ng/mL or higher or abnormal findings on digital rectal examination (DRE)
* Patient with a negative initial urine culture / urinalysis test

Exclusion Criteria:

* Patients who refuses to undergo transperineal prostate biopsy
* Patients who refuses to participate in the research
* Patient who is unable to communicate effectively
* Patient with a documented history of cotrimoxazole allergy
* Patient who has consumed antibiotics for other indications prior to undergoing prostate biopsy
* Patient with urinary tract infection symptoms prior to undergoing prostate biopsy
* Patient with a history of immunodeficiency disorders or long-term corticosteroid use
* Patient with a history of prostate cancer
* Patient with a history of prior prostate biopsy

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2021-07-06 (Actual); Primary Completion 2023-07-06 (Estimated); Study Completion 2023-07-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of infection complications | 24 hours
  The rate of infection complications, including bacteriuria, urinary tract infection (UTI), UTI with fever (febrile UTI), and sepsis, will be measured in both treatment and placebo groups in 24 hours postoperatively.
Incidence of infection complications | 7 days
  The rate of infection complications, including bacteriuria, urinary tract infection (UTI), UTI with fever (febrile UTI), and sepsis, will be measured in both treatment and placebo groups in 7 days postoperatively.
Incidence of infection complications | 14 days
  The rate of infection complications, including bacteriuria, urinary tract infection (UTI), UTI with fever (febrile UTI), and sepsis, will be measured in both treatment and placebo groups in 14 days postoperatively.

SECONDARY OUTCOMES:
Rate of readmission | 7 days
  The rate of readmission will also be assessed in 7 days postoperatively.
Rate of readmission | 14 days
  The rate of readmission will also be assessed in 14 days postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Agus Rizal A. H. Hamid, M.D, Ph.D., Principal Investigator — Universitas Indonesia - Cipto Mangunkusumo Hospital; Harun Wijanarko Kusuma Putra, M.D, B.Med.Sci(Hons), Study Chair — Universitas Indonesia - Cipto Mangunkusumo Hospital; Syamsu Hudaya, M.D., Study Director — Fatmawati General Hospital, Jakarta - Indonesia; Hendy Mirza, M.D., Study Director — Persahabatan Central General Hospital, Jakarta - Indonesia; Dyandra Parikesit, B.Med.Sc., M.D., Study Director — Universitas Indonesia, Depok - Indonesia
Locations (1):
- Dr. Cipto Mangunkusumo Hospital, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No